CLINICAL TRIAL: NCT05745727
Title: A Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Properties of PRX-115 in Adult Volunteers With Elevated Uric Acid Levels.
Brief Title: A Study to Evaluate the Safety, Tolerability, PK, and PD Properties of PRX-115 in Adult Volunteers With Elevated Uric Acid Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PB115-SAD-101
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Gout
Keywords: Uricase; Gout; Uric acid; PRX-115; hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRX-115 (Experimental): Participants will receive a single dose of PRX-115 by IV infusion
  Interventions: Drug: PRX-115
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo by IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRX-115 — Escalating doses of PRX-115 will be given in different cohorts i.e., Cohorts 1 through 8
  Other Names: Escalating doses of PRX-115
  Arms: PRX-115
Drug: Placebo — Escalating doses of Placebo will be given in different cohorts i.e., Cohorts 1 through 8
  Other Names: Placebo to match
  Arms: Placebo

SUMMARY:
This is a Phase 1, double-blind, placebo-controlled, single ascending dose study in participants with elevated uric acid levels. This study will be conducted in approximately 64 adult male and female participants in the dose escalation phase.

DETAILED DESCRIPTION:
Participants will be assigned to 1 of 8 sequential dosing cohorts, each composed of 8 participants (6 active + 2 placebo) who will receive a single dose of PRX-115 or placebo by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 to 65 years of age, inclusive.
2. Serum uric acid greater than 6.0 mg/dL (0.35 mmol/L) at the Screening visit.
3. Body mass index within the range 18.5 to 40 kg/m^2, inclusive, at the Screening visit.
4. Women of childbearing potential may be included only if they have a negative beta human chorionic gonadotropin (β-hCG) test result at Screening.
5. Men and women of childbearing potential and their partners should use double barrier contraception.

Exclusion Criteria:

1. Has any condition known to have arthritis as a clinical manifestation
2. Had greater than or equal to 1 gout flare in the last year prior to either Screening or Day -1.
3. Has clinical evidence of subcutaneous tophi at either Screening or Day -1.
4. Estimated glomerular filtration rate (eGFR) value less than or equal to 60 mL/min/1.73m^2
5. History of significant renal disease, and/or presence of renal stones at either Screening or Day -1.
6. Has a history of anaphylaxis, severe allergic reactions, or severe atopy.
7. History of autoimmune disorders, and/or participant is immunocompromised or treated with immunosuppressive medications.
8. Has evidence of cardiovascular or cerebrovascular disease.
9. History of congestive heart failure, New York Heart Association Class III or IV.
10. BP outside the range of 90 to 150 mm Hg for systolic or 50 to 95 mm Hg for diastolic.
11. Participants with hypertension who are not on stable medication for at least 6 months.
12. Has uncontrolled type 2 diabetes
13. Concurrent treatment with urate lowering drugs (ULDs).
14. Prior exposure to any experimental or marketed uricase (eg, rasburicase [Elitek, Fasturtec], pegloticase [Krystexxa®], pegadricase [SEL-212]).
15. Glucose-6-phosphate dehydrogenase (G6PD) deficiency or known catalase deficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events receiving PRX-115 compared to placebo | Day 0 - Day 85
  To assess the safety and tolerability of a single infusion of PRX-115 as assessed by frequency of drug related adverse events, graded by severity.
Number of participants with abnormal clinically significant clinical laboratory results | Day 0 - Day 85
  Clinical laboratory tests include hematology, coagulation and biochemistry
Number of participants with abnormal clinical vital signs | Day 0 - Day 85
  Vital signs include pulse rate, blood pressure, respiratory rate and tympanic temperature
Number of participants with abnormal clinically significant results from physical examination | Day 0 - Day 85
Number of participants with abnormal clinically significant 12-lead electrocardiogram (ECG) parameters | Day 0 - Day 85

SECONDARY OUTCOMES:
PK of PRX-115: Maximum observed plasma drug concentration (Cmax) | Day 1 - Day 85
  The Cmax PK parameter calculated based on the observed plasma drug concentration versus time curve
PK of PRX-115: Area under the plasma concentration versus time curve (AUC 0-t) | Day 1 - Day 85
  The PK parameter calculated will be Area under the plasma drug concentration-time curve of the last measurable drug concentration (AUC0-t).
PK of PRX-115: Time to maximum observed plasma drug concentration (Tmax) | Day 1 - Day 85
  The PK parameter calculated will be Time to maximum observed plasma drug concentration (T max).
PK of PRX-115: total body clearance (CL) | Day 1 - Day 85
  The PK parameter calculated will be total body clearance (CL).
PK of PRX-115: volume of distribution during the terminal phase (Vd) | Day 1 - Day 85
  The PK parameter calculated will be volume of distribution during the terminal phase (Vd).
PK of PRX-115: Terminal elimination half-life (T ½) | Day 1 - Day 85
  The PK parameter of Terminal elimination half-life (T ½) is calculated based on the plasma drug concentration-time curve
PK of PRX-115: Area under the plasma concentration versus time curve (AUC 0-inf) | Day 1 - Day 85
  The PK parameters calculated will be Area under the plasma drug concentration-time curve from time 0 to infinity (AUC0-inf).
Pharmacodynamics of PRX-115: blood uric acid levels | Day 0 - Day 85
  Pharmacodynamics of PRX-115 by measurement of blood uric acid levels over 85 days
Immunogenicity of PRX-115: measurement of anti-drug antibody levels | Day 1 - Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Mark Marshall, Dr., Principal Investigator — New Zealand Clinical Research
Locations (2):
- New Zealand (2):
  - New Zealand Clinical Research, Grafton, Auckland
  - New Zealand Clinical Research, Christchurch, Christchurch